CLINICAL TRIAL: NCT07315880
Title: Extracellular Fluid Changes During Neoadjuvant Chemotherapy in Breast Cancer: A Prospective Bioimpedance Study
Brief Title: Extracellular Fluid Changes During Neoadjuvant Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Enver Özkurt, Assoc. Prof. Dr., Florence Nightingale Hospital, Istanbul
Other Study IDs: FNH2025-2
Record Dates: First submitted 2025-12-11; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema Arm
Keywords: breast neoplasm; lymphedema; neoadjuvant chemotherapy; breast cancer related lymphedema; extracellular fluid accumulation
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients receiving standard neoadjuvant chemotherapy prior to surgery: This group includes female patients diagnosed with breast cancer who are planned to receive standard neoadjuvant chemotherapy (NACT) prior to any surgical intervention. Participants have not yet undergone breast surgery or axillary lymph node dissection at the time of enrollment. The group will be assessed for early changes in extravascular (extracellular) fluid and subclinical lymphedema using bioimpedance spectroscopy (L-Dex) and arm circumference measurements before and after completion of NACT. All participants follow the same chemotherapy protocol, which may include anthracyclines, cyclophosphamide, paclitaxel, and, if HER2-positive, trastuzumab and pertuzumab.

SUMMARY:
The purpose of this prospective clinical study is to evaluate whether neoadjuvant chemotherapy (NACT) is associated with an increase in extravascular (extracellular) fluid in the ipsilateral upper extremity, an early indicator of breast cancer-related lymphedema (BCRL), in patients with newly diagnosed breast cancer who have not yet undergone breast surgery or axillary lymph node dissection.

Adult patients with a new diagnosis of breast cancer for whom standard NACT is planned will undergo baseline assessments prior to initiation of chemotherapy and follow-up assessments approximately two weeks after completion of NACT. Extravascular fluid status will be evaluated using bioimpedance spectroscopy (L-Dex) and standardized upper extremity circumference measurements.

The primary objective is to assess within-subject changes in extracellular fluid following NACT. Secondary objectives include evaluating the frequency of extracellular fluid increase and exploring associations between extracellular fluid changes and selected patient- and disease-related characteristics, such as age, clinical nodal status, molecular subtype, body mass index, hormone receptor status, and receipt of targeted therapy.

DETAILED DESCRIPTION:
Breast cancer-related lymphedema (BCRL) is a chronic condition that can adversely affect upper extremity function and quality of life. Although BCRL is traditionally regarded as a postoperative complication related to axillary surgery or radiotherapy, accumulating evidence suggests that lymphatic dysfunction and extracellular fluid accumulation may begin earlier in the treatment course, including during neoadjuvant chemotherapy (NACT). Identifying such early, subclinical changes may enable timely preventive strategies.

This prospective, single-center clinical study is designed to evaluate whether neoadjuvant chemotherapy (NACT) is associated with an increase in extravascular (extracellular) fluid in the ipsilateral upper extremity among patients with newly diagnosed breast cancer who have not yet undergone breast surgery or axillary lymph node dissection.

The study was initiated on January 1, 2021, with a planned completion date of December 31, 2025. All participants are recruited and followed at the Istanbul Florence Nightingale Hospital Breast Health Center.

Eligible participants are adult women (≥18 years) with histologically confirmed breast cancer who are scheduled to receive standard NACT. Patients with prior breast or axillary surgery, preexisting clinical lymphedema, incomplete chemotherapy, or non-standard treatment regimens are not included.

Each participant undergoes two standardized assessment visits: a baseline evaluation conducted prior to initiation of NACT and a post-treatment evaluation performed approximately two weeks after completion of NACT and before definitive breast surgery.

At both visits, segmental bioimpedance spectroscopy using the L-Dex U400® device and upper extremity circumference measurements are performed following standardized procedures. For bioimpedance spectroscopy, two consecutive measurements are obtained and averaged to generate the L-Dex score. Arm circumferences are measured at 5-cm intervals along the upper limb, with three measurements averaged at each point. All assessments are conducted by the same trained clinician to ensure measurement consistency.

The standard neoadjuvant chemotherapy regimen consists of four cycles of intravenous doxorubicin (60 mg/m²) and cyclophosphamide (600 mg/m²) administered every 21 days, followed by weekly paclitaxel (80 mg/m²) for 12 weeks. Patients with HER2-positive disease receive trastuzumab and pertuzumab according to standard loading and maintenance dosing schedules concurrently with paclitaxel therapy.

The study evaluates changes in extracellular fluid status using bioimpedance spectroscopy and arm circumference measurements, and explores associations between these changes and selected patient- and disease-related characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older.
* Histologically confirmed diagnosis of breast cancer.
* Planned to receive standard neoadjuvant chemotherapy (NACT) prior to surgery.
* Patients who agreed to participate in the study.
* No contraindications to bioimpedance spectroscopy (BIS), including implanted electronic devices, open wounds or infections on the measurement site, pregnancy, severe non-cancer-related edema, or inability to maintain a supine position during measurement.

Exclusion Criteria:

* Presence of clinically detectable lymphedema at baseline.
* Incomplete or discontinued chemotherapy for any reason.
* Receiving non-standard chemotherapy regimens outside the study protocol.
* Any medical condition or device that prevents accurate BIS measurement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with breast cancer diagnosis
Study Population: The study population includes adult female patients diagnosed with breast cancer who are planned to receive standard neoadjuvant chemotherapy (NACT) prior to any surgical intervention. Participants have not yet undergone breast surgery or axillary lymph node dissection at enrollment. The population includes patients with varying tumor stages and molecular subtypes, including HER2-positive and triple-negative breast cancer. All participants are capable of undergoing bioimpedance spectroscopy (BIS) and arm circumference measurements for the assessment of extravascular fluid changes and subclinical lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Extravascular (Extracellular) Fluid of the Upper Extremity | Baseline (pre-NACT) to two weeks after completion of neoadjuvant chemotherapy
  The primary outcome is the quantitative change in extracellular fluid in the treated upper extremity, measured using bioimpedance spectroscopy (L-Dex U400®) and arm circumference measurements. An increase of ≥6.5 L-Dex units from baseline is considered indicative of subclinical lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Erdoğan İyigün, Prof, Study Chair — Bahçeşehir Üniversitesi
Locations (1):
- Istanbul Florence Nightingale Hospital, Breast Health Center, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
At this time, the plan for sharing individual participant data (IPD) has not been finalized. Decisions regarding data sharing will depend on future considerations, including participant privacy, ethical approvals, and institutional policies.

REFERENCES:
- [Background] Swaroop MN, Ferguson CM, Horick NK, Skolny MN, Miller CL, Jammallo LS, Brunelle CL, O'Toole JA, Isakoff SJ, Specht MC, Taghian AG. Impact of adjuvant taxane-based chemotherapy on development of breast cancer-related lymphedema: results from a large prospective cohort. Breast Cancer Res Treat. 2015 Jun;151(2):393-403. doi: 10.1007/s10549-015-3408-1. Epub 2015 May 5. PMID 25940996
- [Background] Semb KA, Aamdal S, Oian P. Capillary protein leak syndrome appears to explain fluid retention in cancer patients who receive docetaxel treatment. J Clin Oncol. 1998 Oct;16(10):3426-32. doi: 10.1200/JCO.1998.16.10.3426. PMID 9779722
- See also: The Diagnosis and Treatment of Peripheral Lymphedema: 2023 Consensus Document of The International Society of Lymphology — https://pubmed.ncbi.nlm.nih.gov/39207406/
- See also: Impact of adjuvant taxane-based chemotherapy on development of breast cancer-related lymphedema: results from a large prospective cohort — https://pubmed.ncbi.nlm.nih.gov/25940996/
- See also: Evaluation of Long-Term Lymphedema Rate in Patients With Subclinical Lymphedema Diagnosed in the Preoperative Period via Bioimpedance — https://pubmed.ncbi.nlm.nih.gov/39744892/
- See also: L-dex ratio in detecting breast cancer-related lymphedema: reliability, sensitivity, and specificity — https://pubmed.ncbi.nlm.nih.gov/24354107/
- See also: Bioimpedance spectroscopy for breast cancer-related lymphedema assessment: clinical practice guidelines — https://pubmed.ncbi.nlm.nih.gov/36566297/
- See also: Lymphedema following taxane-based chemotherapy in women with early breast cancer — https://pubmed.ncbi.nlm.nih.gov/25411764/
- See also: Treatment factors affecting breast cancer-related lymphedema after systemic chemotherapy and radiotherapy in stage II/III breast cancer patients — https://link.springer.com/article/10.1007/s10549-014-3137-x